CLINICAL TRIAL: NCT07007442
Title: Instrument Assisted Soft Tissue Mobilization Versus Dry Cupping On Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Reda Ahmed Shalby, Bachelor of physiotherapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005096
Record Dates: First submitted 2025-05-25; First posted 2025-06-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intrumented assissted soft tissue mobilization (Experimental): twenty patients Will receive Instrument assisted soft tissue mobilization and Conventional therapy (isometric exercises, stretching, posture correction exercises and cold pack) for 3 sessions per week for 4 weeks
  Interventions: Other: Instrument assisted soft tissue mobilization; Other: conventional therapy
- dry cupping (Experimental): twenty patients Will receive Dry cupping and conventional therapy (isometric exercises, stretching, posture correction exercises and cold pack) for 3 sessions per week for 4 weeks.
  Interventions: Other: dry cupping; Other: conventional therapy
- conventional therapy (Active Comparator): twenty patients will be treated with isometric exercises, stretching, posture correction exercises and cold pack) for 3 sessions per week for 4 weeks.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Instrument assisted soft tissue mobilization — for application of IASTM. the patient will sit on chair in comfortable position, apply lubricant material on treated area (trapezius muscle). Apply IASTM in 30-60 angle for 40 to 120 sec until hyperemia occur for each side+ conventional therapy
  Arms: intrumented assissted soft tissue mobilization
Other: dry cupping — the dry cupping will be aplied by using plastic cups that are placed over localized areas of skin. A vacuum suction is achieved with a manual handheld pump device to create a negative pressure, drawing localized skin and soft tissue structures into the cup+ conventional therapy
  Arms: dry cupping
Other: conventional therapy — the patients will receive Isometric strengthening exercises for cervical Extensors, Flexors, bilateral side Flexors and Rotators (resistance was about 50% of the patient's maximum strength, hold for 10 seconds, for 10 repetitions.Stretching of the upper fibers of trapezius (stretching was held for 30 seconds and repeated 3 times). postural correction exercises in the form of ; 1) Chin tucks exercise is quick and easy to do and it helps strengthening upper thoracic extensors, the muscles that align head over shoulders.2)Corner stretch: provides a deep stretch of the chest and shoulders, which can help maintain good posture.

SUMMARY:
Which is more effective Instrument assisted soft tissue mobilization or Dry cupping on pain intensity, cervical range of motion and functional status in patients with chronic mechanical neck pain?

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal pathology treated by physical therapists around the world. Neck pain is one of the highest complaints in terms of years lived with a disability, increasing the prelevancy of proper management by physical therapists. The overall prevalence of neck pain ranges from 10% to 20%, and the incidence of new neck pain ranging from 10% to 50%. Dry cupping involves the use of glass, plastic or bamboo cups that are placed over localized areas of skin. A vacuum suction is achieved with heat from a flame, a manual handheld pump or electrical pumping devices to create a negative pressure, drawing localized skin and soft tissue structures into the cup . Instrument-assisted soft tissue mobilization (IASTM) is a new technique, which has been known to be effective in reducing muscle tightness in athletes . IASTM is a new tool, which allows clinicians to efficiently locate and treat individuals diagnosed with soft tissue dysfunction .

The use of the instrument is thought to provide a mechanical advantage for the clinician by allowing deeper penetration and more specific treatment, while also reducing imposed stress on the hands

ELIGIBILITY:
Inclusion Criteria:

* 45 patients with chronic mechanical neck pain in the past 3 months.
* Age range from 18 to 35 years old.
* Patients will be from both sexes.
* Body mass index from 18.5 to 24.9 kg/m2.
* Subjects suffer from chronic mechanical neck pain.

Exclusion Criteria:

* Serious injury.
* Tumor.
* Infection.
* Spinal fractures.
* Recent cervical surgery.
* Cervical radiculopathy.
* Skin disease, allergy, hypersensitivity, any malignant or benign tumors.
* Unhealed scars or wounds.
* Pregnancy.
* Known psychiatric condition under treatment or medication.
* Any orthopedic and Neurological condition as cervical PIVD, spondylolisthesis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | up to four weeks
  Visual analogue scale will assess pain intensity.The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale- "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).

SECONDARY OUTCOMES:
Cervical Range of motion | up to four weeks
  The measurements of the cervical range of motion, carried out with the CROM goniometer, The goniometer was placed on the subject's head and a magnetic collar was attached to their shoulders; it was always arranged in the same position with respect to the magnetic pole. During all the measurements, the subjects were seated, with their back straight, and looking ahead; their feet were supported on the floor. The subjects remained in the same sitting position from the moment the recording procedure was started.
  The measurement was performed during "half a cycle" of the movement, i.e., from "the neutral" position to the final range of motion in a given plane.

OTHER OUTCOMES:
neck disability | up to four weeks
  Arabic neck disability index will be used to assess neck disability.The NDI has also been shown to be valid when comparing it to other pain and disability measures. Questions include activities of daily living, such as: personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration and headache. Each question is measured on a scale from 0 (no disability) to 5, and an overall score out of 100 is calculated by adding each item score together and multiplying it by two. A higher NDI score means the greater a patient's perceived disability due to neck pain. The "minimally clinically important change" by patients has been found to be 5 or 10%

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Abdullah, Phd, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Binder AI. Neck pain. BMJ Clin Evid. 2008 Aug 4;2008:1103. PMID 19445809
- See also: Dry Cupping Therapy for Improving Nonspecific Neck Pain and Subcutaneous Hemodynamics — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7384473/